CLINICAL TRIAL: NCT07020689
Title: Combined Airway & Bariatric Surgery (CABS) for Obesity Hypoventilation Syndrome
Brief Title: Transdisciplinary Intervention for Obesity Hypoventilation Syndrome
Acronym: CABS for OHS
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202201000A3; CMRPG1M0101 and CMRPG1M0102 (Other Grant/Funding Number: Chang Gung Medical Foundation)
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2022-08

CONDITIONS: Obesity Hypoventilation Syndrome (OHS); Obstructive Sleep Apnea (OSA)
Keywords: Combined airway and bariatric surgery; Daytime hypercapnia; Obesity hypoventilation syndrome; Obstructive sleep apnea; Sleepiness; Transdisciplinary intervention
MeSH Terms: conditions — Obesity Hypoventilation Syndrome; Sleep Apnea, Obstructive; Sleepiness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obesity with OSA or OHS: Adults aged 20 to 65 years were eligible if they met the following inclusion criteria: (1) BMI ≥ 30 kg/m², and (2) AHI ≥ 5 events/hour. OSA was diagnosed by standard polysomnography. OHS was diagnosed based on the presence of BMI ≥ 30 kg/m², PaCO₂ ≥ 45 mmHg on arterial blood gas (ABG) analysis, and sleep-disordered breathing, following the exclusion of other potential causes of alveolar hypoventilation using pulmonary function tests.
  Interventions: Procedure: CABS

INTERVENTIONS:
Procedure: CABS — Following diagnosis, individuals with OHS were counseled on therapeutic options, including CPAP therapy, body weight reduction, or CABS. The final decision was made through a shared decision-making process. The CABS procedure was conducted under general anesthesia and integrated bariatric and multilevel airway surgery within a single operative session. This transdisciplinary approach aimed to address both sleep-disordered breathing and obesity-related ventilatory compromise. A general surgeon performed the bariatric procedure, while an otorhinolaryngologist conducted the airway surgery sequentially during the same operation. For the bariatric component, laparoscopic sleeve gastrectomy (LSG) was the primary procedure, while laparoscopic Roux-en-Y gastric bypass was reserved for individuals with significant gastroesophageal reflux or poorly controlled diabetes. Airway surgery encompassed interventions at the nasal, palatal, and lingual levels.

SUMMARY:
The aims of this prospective observational cohort study are threefold: (1) to assess the prevalence of obesity hypoventilation syndrome (OHS) in individuals with obesity and obstructive sleep apnea (OSA) and identify associated risk factors, (2) to determine clinical predictors of OHS, and (3) to evaluate the therapeutic outcomes of combined airway and bariatric surgery (CABS) in this population.

DETAILED DESCRIPTION:
This study was approved by the Institutional Review Board of Chang Gung Medical Foundation on August 8, 2022 (IRB No. 202201000A3). Written informed consent was obtained from all participants. All procedures adhered to the principles outlined in the Declaration of Helsinki and were reported in accordance with the Strengthening the Reporting of Observational Studies in Epidemiology (STROCSS) guidelines.

This was a two-year prospective observational cohort study conducted at the tertiary referral sleep center of Linkou Chang Gung Memorial Hospital from December 1, 2022, to November 30, 2024. Obesity hypoventilation syndrome (OHS) was diagnosed based on the presence of BMI ≥ 30 kg/m², PaCO₂ ≥ 45 mmHg on arterial blood gas (ABG) analysis, and sleep-disordered breathing, following the exclusion of other potential causes of alveolar hypoventilation using pulmonary function tests.

Adults aged 20 to 65 years were eligible if they met the following inclusion criteria: (1) BMI ≥ 30 kg/m², and (2) AHI ≥ 5 events/hour. Individuals were excluded if they had (1) persistent decompensated hypercapnic respiratory failure (arterial pH < 7.3), (2) acute respiratory failure requiring invasive mechanical ventilation, (3) significant neuromuscular disease, chest wall deformities, or pulmonary disease contributing to hypoventilation, (4) unstable coronary artery disease, or (5) cognitive impairment precluding informed consent or protocol adherence.

Following diagnosis, individuals with OHS were counseled on therapeutic options, including continuous positive airway pressure (CPAP) therapy, body weight reduction, or combined airway and bariatric surgery (CABS). The final decision was made through a shared decision-making process.

Outcome measures included (1) Polysomnography: All participants underwent attended level I polysomnography using the Nicolet UltraSom System (Nicolet, Madison, WI). AHI was the primary sleep parameter, defined as the total number of apneas (≥ 90% airflow reduction for ≥10 seconds) and hypopneas (> 50% airflow reduction with ≥ 3% oxygen desaturation or arousal) per hour of sleep. Scoring was performed by a single blinded sleep specialist. (2) Pulmonary function testing: Spirometry was performed using a handheld spirometer in accordance with international guidelines. Parameters included forced vital capacity (FVC), forced expiratory volume in 1 second (FEV₁), and FEV₁/FVC ratio. (3) Gas exchange: ABG analysis was conducted during daytime hours with the participant seated and breathing room air after resting for at least 60 minutes. (4) Epworth sleepiness scale: Daytime sleepiness was assessed using the Epworth Sleepiness Scale (ESS), a validated 8-item questionnaire with total scores ranging from 0 to 24; higher scores indicate greater daytime sleepiness.

The prevalence of OHS was calculated as the proportion of individuals diagnosed with OHS among those with concurrent obesity and obstructive sleep apnea (OSA). A multivariate logistic regression analysis with forward selection was conducted to identify independent predictors of OHS. Receiver operating characteristic (ROC) curve analysis was used to determine the optimal cut-off points for various predictors. To evaluate the effects of the CABS intervention, pre- and post-operative changes in clinical parameters were compared.

ELIGIBILITY:
Inclusion Criteria:

(1) BMI ≥ 30 kg/m², and (2) AHI ≥ 5 events/hour.

Exclusion Criteria:

(1) persistent decompensated hypercapnic respiratory failure (arterial pH < 7.3), (2) acute respiratory failure requiring invasive mechanical ventilation, (3) significant neuromuscular disease, chest wall deformities, or pulmonary disease contributing to hypoventilation, (4) unstable coronary artery disease, or (5) cognitive impairment precluding informed consent or protocol adherence.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study enrolled consecutive patients with obesity and OSA at the tertiary referral sleep center of Linkou Chang Gung Memorial Hospital from September 1, 2022, to August 31, 2024. OHS was diagnosed based on the presence of BMI ≥ 30 kg/m², PaCO₂ ≥ 45 mmHg on ABG analysis, and sleep-disordered breathing, following the exclusion of other potential causes of alveolar hypoventilation using pulmonary function tests.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
AHI | From enrollment to the end of treatment at 12 months.
  All participants underwent attended level I polysomnography using the Nicolet UltraSom System (Nicolet, Madison, WI). Apnea-hypopnea index (AHI) was the primary sleep parameter, defined as the total number of apneas (≥ 90% airflow reduction for ≥10 seconds) and hypopneas (> 50% airflow reduction with ≥ 3% oxygen desaturation or arousal) per hour of sleep. Scoring was performed by a single blinded sleep specialist.

SECONDARY OUTCOMES:
FEV₁/FVC ratio | From enrollment to the end of treatment at 12 months.
  Spirometry was performed using a handheld spirometer in accordance with international guidelines. Parameters included forced vital capacity (FVC), forced expiratory volume in 1 second (FEV₁), and FEV₁/FVC ratio.
PaCO₂ | From enrollment to the end of treatment at 12 months
  Arterial blood gas (ABG) analysis was conducted during daytime hours with the participant seated and breathing room air after resting for at least 60 minutes.
ESS score | From enrollment to the end of treatment at 12 months.
  Daytime sleepiness was assessed using the Epworth Sleepiness Scale (ESS), a validated 8-item questionnaire with total scores ranging from 0 to 24; higher scores indicate greater daytime sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Hsueh-Yu Li, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of ENT, Linkou Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baird K, Comis LE, Joe GO, Steinberg SM, Hakim FT, Rose JJ, Mitchell SA, Pavletic SZ, Figg WD, Yao L, Flanders KC, Takebe N, Sarantopoulos S, Booher S, Cowen EW. Imatinib mesylate for the treatment of steroid-refractory sclerotic-type cutaneous chronic graft-versus-host disease. Biol Blood Marrow Transplant. 2015 Jun;21(6):1083-90. doi: 10.1016/j.bbmt.2015.03.006. Epub 2015 Mar 12. PMID 25771402